CLINICAL TRIAL: NCT00864019
Title: A Single-Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalence Study of Sertraline 100 mg Tablets Under Fed Conditions
Brief Title: A Relative Bioavailability Study of Sertraline HCl 100 mg Tablets Under Non-fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 20-683-1G
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Sertraline; Healthy subjects
MeSH Terms: interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Sertraline HCl 100 mg tablets, single dose
  Interventions: Drug: Sertraline HCl 100 mg tablets, single dose
- B (Active Comparator): Zoloft® 100 mg tablets, single dose
  Interventions: Drug: Zoloft® 100 mg tablets, single dose

INTERVENTIONS:
Drug: Sertraline HCl 100 mg tablets, single dose — A: Experimental SSubjects received Purepac formulated products under non-fasting conditions
  Other Names: Sertraline
  Arms: A
Drug: Zoloft® 100 mg tablets, single dose — B: Active comparator Subjects received Pfizer formulated products under non-fasting conditions
  Other Names: Sertraline
  Arms: B

SUMMARY:
To compare the rate of absorption and oral bioavailability of a test formulation of Sertraline 100 mg tablets manufactured by Purepac Pharmaceutical Company to an equivalent oral dose of the commercially available reference product, Zoloft® manufactured by Pfizer Inc. Following an overnight fast of at least 10 hours, subjects will consume a standard high-calorie, high-fat breakfast meal. This standard breakfast will begin 30 minutes prior to each dose.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: A single-dose, open-label, randomized, two-period crossover study

Official Title: A Single-Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalence Study of Sertraline 100 mg Tablets Under Fed Conditions

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a male or non-pregnant, non-breast-feeding female.
* Subject must be between 18 and 55 years of age inclusive.
* Subject's body weight should be within ±15% of the ideal body weight for their height and estimated frame based on the Metropolitan Life Insurance Company Table.
* Female subjects --- not surgically sterile or at least two years postmenopausal --- must agree to utilize one of the following forms of contraception, if sexually active with a male partner, from screening through completion of the study. Approved forms of contraception are abstinence, hormonal (oral, implant, transdermal or injection), double barrier (condom and diaphragm with spermicide), IUD, or vasectomized partner (6 months minimum).
* Subject must voluntarily consent to participate in this study and provide their written informed consent prior to completion of any study-specific procedures.
* Subject is willing and able to remain in the study unit for the entire duration of each confinement period and return to the study site for all out-patient visits.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic or psychiatric disease or any other condition which, in the opinion of the Investigator would jeopardize the safety of the subject or the validity of the study results.
* Has a clinically significant abnormal finding on the physical exam, medical history or clinical laboratory results at screening.
* History or presence of allergic or adverse response to the study drug or related drugs.
* Has been on a significantly abnormal diet during the four weeks preceding the first dose of study medication.
* Has donated blood or plasma within 30 days prior to the first dose of study medication.
* Has participated in another clinical trial within 30 days prior to first dose of study medication.
* Has used any over-the-counter (OTC) medication including vitamins, within 7 days prior to the first dose of study medication.
* Has used any prescription medication, except hormonal contraceptive or hormonal replacement therapy, within 7 days prior to the first dose of study medication.
* Has been treated with any known enzyme altering drugs such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication.
* Has smoked or used tobacco products within 60 days prior to the first dose of study medication.
* Female with a positive pregnancy test.
* Positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates).
* Has had a positive test for, or has been treated for hepatitis B, hepatitis C or HIV.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-08; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Daniel V. Freeland,, D.O., CCI, Principal Investigator — CEDRA Clinical Research, LLC
Locations (1):
- CEDRA Clinical Research, LLC, Austin, Texas, United States